CLINICAL TRIAL: NCT00868920
Title: A Phase IV, Randomized, Double-Blind, Controlled Study of the Effects of Patient-Controlled Sedation vs. Anesthesiologist-Administered Sedation With Propofol and Remifentanil on Rate of Disordered Breathing in Subjects Undergoing Elective Colonoscopy
Brief Title: Patient-Controlled Sedation Versus Anesthesiologist-Administered Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 806514
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The Graseby 3300 PCA pump will be loaded with a mixture of propofol 10 mg/cc containing 10 µg/cc remifentanil. The loading and demand doses will be individualized based on patient weight, height, age, and gender.
  The initial loading phase of sedation will be performed by the anesthesiologist to permit estimation of patient sensitivity. Following the initial loading dose, a series of button presses will be issued by the anesthesiologist to achieve a state of moderate sedation, as determined by a decrease in BIS to the range of 75-80. Once this state has been reached, the button will be transferred to the patient for Patient C0ntrolled Sedation.
  Interventions: Other: patient control of pump
- 2 (Experimental): The Graseby 3300 PCA pump will be loaded with a mixture of propofol 10 mg/cc containing 10 µg/cc remifentanil. The loading and demand doses will be individualized based on patient weight, height, age, and gender.
  The initial loading phase of sedation will be performed by the anesthesiologist to permit estimation of patient sensitivity. Following the initial loading dose, a series of button presses will be issued by the anesthesiologist to achieve a state of moderate sedation, as determined by a decrease in BIS to the range of 75-80. Once this state has been reached,the anesthesiologist will control the sedation.
  Interventions: Other: anesthesiologist controlled sedation

INTERVENTIONS:
Other: patient control of pump — Patient controls sedation pump during colonoscopy.
  Arms: 1
Other: anesthesiologist controlled sedation — Anesthesiologist will control the sedation pump during colonoscopy.
  Arms: 2

SUMMARY:
The purpose of this study is to see whether patients controlling their own sedation during colonoscopy are less likely to need help breathing than when an anesthesiologist controls the medicine, and whether we can predict when the need for help will occur. The pump used in the study is approved for clinical use by the FDA, as are the medicines used in the pump.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective, outpatient colonoscopy
2. Age ≥ 18, <90
3. Meet criteria for conscious sedation (HUP Policy 1-12-11, Appendix F), as determined by the attending gastroenterologist and confirmed by the anesthesiologist by review of history
4. Able to give informed consent

Exclusion Criteria:

1. Have a history of allergy or adverse reaction to propofol or remifentanil
2. Have a condition which would pose an elevated risk for administration of propofol, including primary hyperlipoproteinemia, diabetic hyperlipemia, and pancreatitis.
3. Female of child-bearing potential (under 50 without surgical sterilization)
4. Unable to understand the use of Patient Contolled Sedation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the depth of sedation, | during colonoscopy procedure

SECONDARY OUTCOMES:
The secondary outcome measure is rate of respiratory depression | during colonoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jeff E Mandel, MD MS, Principal Investigator — University of Pennsylvania, Anesthesia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mandel JE, Lichtenstein GR, Metz DC, Ginsberg GG, Kochman ML. A prospective, randomized, comparative trial evaluating respiratory depression during patient-controlled versus anesthesiologist-administered propofol-remifentanil sedation for elective colonoscopy. Gastrointest Endosc. 2010 Jul;72(1):112-7. doi: 10.1016/j.gie.2010.01.031. Epub 2010 May 20. PMID 20493481